CLINICAL TRIAL: NCT03782701
Title: The Effect of Lumify™ (Brimonidine Tartrate Ophthalmic Solution 0.025%) on Palpebral Fissure Height
Brief Title: The Effect of Lumify™ Eyedrops on Eyelid Position
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Wendy Lee, Associate Professor of Ophthalmology and Dermatology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180895
Record Dates: First submitted 2018-11-12; First posted 2018-12-20 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Eyelid Droop
MeSH Terms: conditions — Blepharoptosis | interventions — Brimonidine Tartrate

STUDY DESIGN:
Intervention Model Description: The left and right eye of each subject will be randomized to receive either Lumify or balanced saline placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lumify Eye Drop (Active Comparator): Participants will be randomized to receive a single drop of Lumify to either the left or right eye.
  Interventions: Drug: Brimonidine tartrate ophthalmic solution 0.025%
- Saline Solution Eye Drop (Active Comparator): Participants will be randomized to receive a single drop of sterile balanced saline solution to either the left or right eye.
  Interventions: Other: Sterile balanced saline solution

INTERVENTIONS:
Drug: Brimonidine tartrate ophthalmic solution 0.025% — One time dosing of brimonidine tartrate ophthalmic solution 0.025% (1 drop applied to ocular surface)
  Other Names: Lumify
  Arms: Lumify Eye Drop
Other: Sterile balanced saline solution — One time dosing of sterile balanced saline solution (1 drop applied to ocular surface)
  Arms: Saline Solution Eye Drop

SUMMARY:
The purpose of the research is to see if Lumify™ has an effect on eyelid position.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and above able to provide informed consent to participate
* Subject with stable ocular health, defined as no ocular conditions requiring ongoing topical therapy or recent surgical intervention

Exclusion Criteria:

* Adults unable to consent
* Prisoners
* Pregnant women.
* Known contradictions or sensitivities to study medication (brimonidine)
* Ocular surgery within the past 3 months or refractive surgery within the past six months
* Grossly abnormal lid margins, anatomical abnormalities, previous eyelid or orbital surgery
* Variable ptosis or eyelid position (e.g., myasthenia gravis, thyroid eye disease, or blepharospasm)
* Significant pre-existing ptosis of any cause (defined as margin reflex distance 1 < 1mm)
* Any ocular or systemic condition that, in the opinion of the investigator, would confound study data, interfere with the subject's study participation, or affected the subject's safety or trial parameters
* Presence of an active ocular infection
* Prior (within 5 days of beginning study treatment) use of eye whiteners (eg, vasoconstrictors), decongestants, antihistamines (including over the counter and herbal topical ophthalmic medications), phenylephrine dilating drops, any other topical ophthalmic agents
* Inability to sit comfortably for 15 - 30 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy W Lee, MD, MS, Principal Investigator — Bascom Palmer Eye Institute
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eye
Groups:
- All Participants: All participants received both the Lumify and saline solution. The left and right eye of each subject was randomized to receive either Lumify or balanced saline solution.
Period: Overall Study
Arm/Group | All Participants
Started | 43; 86 eye
Lumify | 43; 43 eye
Saline Solution | 43; 43 eye
Completed | 43; 86 eye
Not Completed | 0; 0 eye

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Palpebral Fissure Height
Description: Objective measurement of distance between inner margin of upper and lower eyelids from clinical photographs.
Time Frame: Baseline, 5, 15 and 30 minutes after application
Population: All participants received both the Lumify and saline solution. The left and right eye of each subject was randomized to receive either Lumify or balanced saline solution. Measurements from 3 participants were not collected due to brow ptosis.
Measure: Mean (Standard Deviation); unit: milimeter
Units Other Than Participants: eye
Arm/Group | Lumify Eye Drop | Saline Solution Eye Drop
Number analyzed (Participants) | 40 | 40
Number analyzed (eye) | 40 | 40
milimeter
  Baseline | 9.64 (1.71) | 9.66 (1.62)
  5 minutes after application | 9.92 (1.33) | 9.96 (1.35)
  15 minutes after application | 9.85 (1.42) | 9.96 (1.40)
  30 minutes after application | 9.86 (1.32) | 9.84 (1.26)

2. Secondary Outcome: Intraocular Pressure
Description: Measurement of intraocular pressure using handheld Tono-Pen(tm) tonometer
Time Frame: Baseline, 5, 15 and 30 minutes after application
Population: All participants received both the Lumify and saline solution. The left and right eye of each subject was randomized to receive either Lumify or balanced saline solution. Intraocular Pressure was only conducted at Baseline and 30 minutes post application.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eye
Arm/Group | Lumify Eye Drop | Saline Solution Eye Drop
Number analyzed (Participants) | 43 | 43
Number analyzed (eye) | 43 | 43
mmHg
  Baseline | 16.54 (3.63) | 16.70 (3.42)
  30 minutes after applciation | 15.54 (3.30) | 15.58 (2.99)

3. Secondary Outcome: Eye Redness
Description: Eye redness will be reported as the number of participants achieving a score of ocular redness from clinical photographs as 0 (none), 1 (mild), 2 (moderate) and 3 (severe).
Time Frame: Baseline, 5, 15 and 30 minutes after application
Population: All participants received both the Lumify and saline solution. The left and right eye of each subject was randomized to receive either Lumify or balanced saline solution.
Measure: Count of Participants; unit: Participants
Arm/Group | Lumify Eye Drop | Saline Solution Eye Drop
Number analyzed (Participants) | 43 | 43
Participants
  Baseline - None | 24 | 25
  Baseline - Mild | 17 | 16
  Baseline - Moderate | 2 | 2
  Baseline - Severe | 0 | 0
  5 minutes after application - None | 38 | 6
  5 minutes after application - Mild | 4 | 19
  5 minutes after application - Moderate | 1 | 17
  5 minutes after application - Severe | 0 | 1
  15 minutes after application - None | 40 | 18
  15 minutes after application - Mild | 2 | 24
  15 minutes after application - Moderate | 1 | 1
  15 minutes after application - Severe | 0 | 0
  30 minutes after application - None | 41 | 26
  30 minutes after application - Mild | 1 | 17
  30 minutes after application - Moderate | 1 | 0
  30 minutes after application - Severe | 0 | 0

4. Secondary Outcome: Eye Discomfort
Description: Eye discomfort will be reported as the number of participants reporting subjective ocular discomfort score from 0 (none), 1 (mild), 2 (mild) and 3 (severe).
Time Frame: Baseline, 5, 15 and 30 minutes after application
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lumify Eye Drop | Saline Solution Eye Drop
Number analyzed (Participants) | 43 | 43
Participants
  Baseline - None | 43 | 43
  Baseline - Mild | 0 | 0
  Baseline - Moderate | 0 | 0
  Baseline - Severe | 0 | 0
  5 minutes after application - none | 40 | 38
  5 minutes after application - mild | 3 | 4
  5 minutes after application - moderate | 0 | 0
  5 minutes after application - severe | 0 | 1
  15 minutes after application - none | 41 | 40
  15 minutes after application - mild | 1 | 2
  15 minutes after application - moderate | 1 | 1
  15 minutes after application - severe | 0 | 0
  30 minutes after application - none | 39 | 40
  30 minutes after application - mild | 4 | 3
  30 minutes after application - moderate | 0 | 0
  30 minutes after application - severe | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 minutes
Arm/Group | Lumify Eye Drop | Saline Solution Eye Drop
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 6/43 | 2/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumify Eye Drop (N=43) | Saline Solution Eye Drop (N=43)
Eye Pain (Eye disorders) | 2 (2) | 2 (2)
Eye Itchiness (Eye disorders) | 1 (1) | 0 (0)
Eye Dryness (Eye disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT03782701/Prot_SAP_001.pdf